CLINICAL TRIAL: NCT03952052
Title: Detection by Digital PCR and Next Generation Sequencing of Recurrent Mutations in Waldenström's Disease and Study of Their Distribution in the Different Biological Compartments
Brief Title: Detection of Recurrent Mutations in Waldenström's Disease
Acronym: DigiWAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB 18.06
Record Dates: First submitted 2019-05-07; First posted 2019-05-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Waldenstrom's Disease
Keywords: MRD; Mutation; Next Generation sequencing; Digital Polymeras Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient enrolled (Other): Recurrent mutations determination
  Interventions: Other: Determination of mutation

INTERVENTIONS:
Other: Determination of mutation — Recurrent mutation determination by digital PCR and next generation sequencing

SUMMARY:
Waldenström's disease (WM) is a rare, low-grade lymphoid hematopathy, accounting for 1 to 2% of malignant hematopathies and mainly affecting the elderly. This disease is characterized by lymphoplasmocyte cells infiltration into the bone marrow and by the production of a monoclonal IgM protein in the serum. This disease is accompanied by clinical manifestations of hepato-splenomegaly, signs of hyperviscosity, peripheral neuropathies and biological signs with the presence of cytopenias and cryoglobulinemia. Some forms present node or splenic involvement. While the asymptomatic form maintains overall survival close to that of the healthy subject, the symptomatic form is subject to frequent relapses and remains incurable.

Current recommendations for the diagnosis and monitoring of this disease are based on protein electrophoresis from a blood sample to quantify monoclonal IgM production and a myelogram or bone marrow biopsy showing medullary infiltration by lymphoplasmocytic cells. However, protein electrophoresis is an imprecise examination since it does not quantify tumour B lymphocytes and has limitations, particularly in the case of poorly secreting forms.

More than 90% of Waldenström cases have the L265P mutation of the MYD88 gene. Although this mutation is not found only in these diseases, it can help in the diagnosis. Other mutations are also present in this pathology. These mutations can define prognostic factors or possibly make it possible to identify therapeutic targets.

The development of new technologies makes it possible, on the one hand, to follow the L265P mutation of MYD88 over time as a marker of response to treatment and, on the other hand, to define these prognostic markers or therapeutic targets.

This study will first determine the best method for monitoring the mutation of MYD88. In a second step, the investigators will evaluate the best type of sampling and in particular whether this mutation is present in the blood in order to limit the invasive procedures such as bone marrow sampling can be limited. Finally, the investigators will evaluate the prognostic

DETAILED DESCRIPTION:
The L265P mutation of MYD88 appears as an early oncogenic event in the occurrence of Waldenström disease and may already be present at the Monoclonal Gammapathy of Undetermined Signification (MGUS) to IgM stage suggesting a continuum between the two stages of the disease. The determination of IgM as a marker of the disease has limits since it does not allow direct quantification of the clonal population and is taken failing this in the case of poorly secreting forms. Monitoring the L265P mutation of MYD88 as a marker of minimal residual disease therefore appears to be a biomarker of major interest in these diseases. The kinetics of this marker particularly during treatment could allow to modify the therapeutic management of patients at an early stage and to assess the risk of resistance to treatment.

Several published studies show the interest of monitoring the L265P mutation of MYD88 in MW in particular by quantification of the mutation by allele-specific PCR. The detection limit studied was 0.1%. The recent development of new techniques and in particular digital PCR makes it possible to obtain lower detection thresholds that could be more compatible with the notion of minimal residual disease monitoring.

The originality of this study is based on the comparison of the quantification of the MYD88 L265P mutation in all affected biological compartments (blood, plasma, bone marrow or CD19+ cells) but especially in the monitoring of the mutation at two points of minimal residual disease (mid-treatment and end of treatment).

One of the parts of the project is the study of the allelic frequency of the L265P mutation of the MYD88 gene in circulating tumor DNA (ctDNA). It has been shown in many pathologies and in particular in other B lymphocytic hematologies such as Hodgkin's lymphoma or diffuse large cell B lymphoma, that mutations present at the tumor level could be found in circulating tumor DNA. Analysis of free tumor DNA circulating in patients' plasma can therefore be used to characterize the disease at the molecular level with a less invasive sample than myelogram or bone marrow biopsies. The search for other associated mutations also reinforces the originality of the project. These combined data must be able to lead to changes in the clinical management of patients.

In this study, the allele frequency of the L265P mutation of MYD88 will be compared . by 3 different techniques: specific allele PCR, digital PCR and new generation sequencing. In this way, investigators will evaluate the technique that has the best sensitivity and specificity to be used as a marker for residual disease. These data will be compared to the reference technique, protein electrophoresis. This evaluation will be conducted in total mononuclear cells, DNAct, marrow and CD19+ sorted cells. Then, the investigators will follow the kinetics of this mutation during the treatment at two points : mid-treatment and end of treatment.

Characterization of the mutation profile of these tumors allows prognostic factors to be defined and may identify potential new therapeutic targets. This study will be realised by new generation sequencing. Some of genes with mutations involved in treatment resistance will be studied such as CXCR4. The mutations of CXCR4 are involved in the resistance to ibrutinib. ARID1A mutations are also found in 20% of cases as well as TP53, KMT2D, CD79B, MYBBP1A mutations.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* recently diagnosed for Waldenström's disease
* not yet treated for Waldenström's disease

Exclusion Criteria:

* Pregnancy or breast feeding
* HBV or HBC positive
* HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Quantification of MYD88 L265P mutation | one year
  Comparison of level of MYD88L265P mutationin different biological compartment c.

SECONDARY OUTCOMES:
Allelic frequency of L265P mutation of MYD 88 gene | one year
  Comparison of allelic frequency determined by three different techniques (next generation sequencing, digital PCR and specific allele PCR)
Kinetics of mutation | one year
  determination of the kinetics of mutation

CONTACTS AND LOCATIONS:
Overall Officials: Pascaline Etancelin, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No